CLINICAL TRIAL: NCT05372172
Title: Tennessee Alzheimer's Project
Acronym: TAP
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Angela Jefferson, Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: 211309; P20AG068082 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-05-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Aging; Alzheimer Disease; Biomarker; Cognitive Dysfunction; Mild Cognitive Impairment; Dementia; Cognition
Keywords: Alzheimer's disease; biomarkers; brain MRI; mild cognitive impairment; vascular risk factors; longitudinal studies
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebral spinal fluid, plasma, serum, PAXGene, blood clot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cognitively unimpaired: A consensus team determined cognitive status according to the National Institute on Aging and Alzheimer's Association Workgroup guidelines.
  Interventions: Other: none, observational study
- Mild cognitive impairment: A consensus team determined cognitive status according to the National Institute on Aging and Alzheimer's Association Workgroup guidelines.
  Interventions: Other: none, observational study
- Alzheimer's disease: A consensus team determined cognitive status according to the National Institute on Aging and Alzheimer's Association Workgroup guidelines.
  Interventions: Other: none, observational study

INTERVENTIONS:
Other: none, observational study — none, observational study

SUMMARY:
The primary objective of the Vanderbilt Alzheimer's Disease Research Center (VADRC) is to provide local and national researchers with access to a well-characterized and diverse clinical cohort, including participant referrals, biosamples, clinical data, and neuroimaging data. The VADRC Clinical Core will create an infrastructure to support research efforts of both local and national investigator studies to develop early detection, prevention, and treatment strategies for Alzheimer's disease. The Clinical Core intends to enroll up to 1000 participants, including individuals who are cognitively unimpaired, have mild cognitive impairment, or have Alzheimer's disease. This cohort of about 1000 participants will be called the Tennessee Alzheimer's Project. Participants will be seen annually for comprehensive clinical characterization and then referred to other studies to enhance Alzheimer's disease research activities.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a growing public health crisis affecting 5.8 million Americans. With the aging population, AD prevalence is expected to double by 2040. Successful AD prevention and effective therapies require distilling complexities of the disease to better model disease onset, progression, and treatment response. The purpose of the Vanderbilt Alzheimer's Disease Research Center (VADRC) is to provide a better understanding of AD and related dementias, and to serve as the institutional hub of clinical, research, and educational initiatives in AD. The Center will play an essential role in expanding AD discoveries and reducing the burden of AD locally and nationally. To do so, the VADRC will support multiple human studies and model systems research over the coming years. For the Tennessee Alzheimer's Project, the team will establish, phenotype, and annually follow a cohort of adults age 60 and older with and without memory problems. Phenotyping will include standardized protocols implemented across the entire national ADRC network as part of the National Alzheimer's Coordinating Center as well as protocols specific to our local site, including (but not limited to) venous blood draw, questionnaires, physical examination, echocardiogram, neuropsychological assessment, multi-modal neuroimaging, and cerebrospinal fluid acquisition via lumbar puncture. As part of the Center's autopsy program, the investigators will ask all Tennessee Alzheimer's Project participants to consider post-mortem donation of their brain, eyes, and a small skin sample. While fluid and neuroimaging biomarkers exist for some neuropathologies associated with AD and related dementias, postmortem characterization is the only current way to definitively confirm the presence and severity of disease. Locally, a robust tissue bank with excellent ante-mortem phenotyping will provide invaluable tissue for analyses distilling the complexities of AD.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Meet standard criteria for (a) cognitively unimpaired, (b) mild cognitive impairment, or (c) Alzheimer's disease
* English speaking
* Individuals who lack decisional capacity to provide informed consent at baseline will not be enrolled in the study

Exclusion Criteria:

* No available reliable study partner (reliable is defined as someone who interacts significantly with the participant and is available to participate in study visits in person or by phone)
* History of major psychiatric illness (e.g., schizophrenia, bipolar), neurological illness (e.g., epilepsy, multiple sclerosis, Parkinson's disease), or head injury with significant loss of consciousness.
* Unable to undergo MRI (e.g., claustrophobia, ferrous metal in body)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive status | baseline to year 3
  Change in cognitive status assessed by the Uniform Dataset according to the National Institute on Aging and Alzheimer's Association Workgroup guidelines determined by a consensus team.
APOE Genotype | baseline to year 3
  APOE e4 allele status
White matter hyperintensities Volume | baseline to year three
  White matter lesion volume measured by FLAIR imaging modality
Grey Matter Volume | baseline to year three
  Grey matter volume measured by T1 imaging modality
Cerebral Blood Flow | baseline to year three
  Resting cerebral blood flow to brain regions measured by T3 perfusion
Lacunar infarcts | baseline to year three
  Number of lacunar infarcts measured by MRI
Microbleeds | baseline to year three
  Number of microbleeds measured by MRI
Left ventricular ejection fraction | baseline to year three
  Left ventricular ejection fraction measured by echocardiogram
Cardiac output | baseline to year three
  Amount of blood the heart pumps from each ventricle per minute (litres per minute (L/min)), measured by echocardiogram
Stroke volume | baseline to year three
  Stroke volume measured by echocardiogram
Heart rate | baseline to year three
  Heart rate measured by echocardiogram
Biological markers for Alzheimer's disease | baseline to year three
  Tau, amyloid, and neurodegenerative levels in cerebrospinal fluid samples
Blood based biological marker for Alzheimer's disease | baseline to year three
  Tau, amyloid, and neurodegenerative levels in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Angela Jefferson, PhD, Principal Investigator — Professor of Neurology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No